CLINICAL TRIAL: NCT01222013
Title: Phase II Study for Safety and Efficacy Evaluation of Imatinib Mesylate in Children With Acute Lymphoblastic Leukemia (ALL) Philadelphia Chromosome-positive (Ph+)
Brief Title: Study for Safety and Efficacy Evaluation of Imatinib Mesylate in Children With Acute Lymphoblastic Leukemia (ALL) Philadelphia Chromosome-positive (Ph+)
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was suspended before recruitment, due to logistic issues.
Sponsor: Renato Melaragno (Other)
Responsible Party: Sponsor-Investigator, Renato Melaragno, MD, Hospital Santa Marcelina
Organization: Hospital Santa Marcelina (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571ABR22T
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Acute Lymphoblastic Leukemia (ALL) Philadelphia Chromosome-positive (Ph+)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib Mesylate (Experimental)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — patient will receive Imatinib (Glivec®), 300 mg/m²/day, per oral, in conjunction with chemotherapy, maximum dose allowed 400 mg/dia.
  Other Names: Glivec, MI

SUMMARY:
The purpose of this study is to evaluate the efficacy, through molecular response and event-free survival, about the use of Imatinib in conjunction with chemotherapy after BFM "like" Induction in children with ALL Ph+.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose: therapy-naïve ALL, except for patients that performed Induction for ALL (33 days) exactly as this protocol and; documented Ph+, to be confirmed by conventional cytogenetic - t(9;22) (q34;q11) or FISH and/or gene BCR-ABL presence by RT-PCR or FISH.
2. Female patients of childbearing age, should have pregnancy test (blood βhCG) performed before treatment initiation. Effective contraception must be used during treatment. Pregnant women won't be included.
3. Life expectation > 8 weeks.
4. Medications: antineoplastic treatment-naïve, including corticotherapy, except for patients that performed Induction for ALL (33 days) exactly as this protocol.
5. Signed ICF by child legal responsible.
6. Laboratory: renal function (serum creatinine ≤ 1,5 x ULN and/or Clearance ≥70 ml/min/1,73m2), hepatic function (total bilirubin ≤ 1,5 x ULN, TGP/TGO < 10 x ULN and albumin > 2 g/dl.

Exclusion Criteria:

1. Any inclusion criteria missing.
2. Pregnant patient or breastfeeding.
3. Patient considered incapable to follow purposed treatment.
4. Subject with infectious process, in activity, grade IV.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy, through molecular response and event-free survival, about the use of Imatinib in conjunction with chemotherapy after BFM "like" Induction in children with ALL Ph+. | Up to 24 months.
  Cytogenetic and molecular response will be evaluate at the end of Induction I (D33), before each consolidation block (HR 1, 2 and 3), before re-induction, before maintenanceand at the end of therapy.

SECONDARY OUTCOMES:
Evaluate toxicity and tolerability in the administration of Imatinib in conjunction with chemotherapy in children with ALL Ph+. | Up to 24 months
  Toxicity and tolerability will be verified in every visit according through:
  * Adverse events during the study.
  * Laboratory exams.
  * Vital signs and body weight.
  * Physical evaluation.
  * Concomitant medication.